CLINICAL TRIAL: NCT01391650
Title: Rotational and Anteroposterior Stability of the Knee Joint After Single- and Double- Bundle ACL Reconstruction
Brief Title: Stability of the Knee Joint After Single and Double Bundle Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Znojmo (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Komzak Martin, M.D., proncipal investigator, Hospital Znojmo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DBVSB
Record Dates: First submitted 2011-05-20; First posted 2011-07-12 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: ACL; double-bundle; navigation system
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- biomechanic of the knee (Experimental)
  Interventions: Procedure: 'biomechanic of the knee'

INTERVENTIONS:
Procedure: 'biomechanic of the knee' — 20 patients had their ACL replaced by SB reconstruction from hamstrings, 20 patients double - bundle technique with AM bundle being reconstructed first, and 20 patients with the PL bundle first.
  Other Names: replacement of ACL

SUMMARY:
The purpose of this prospective study is to evaluate the influence of both bundles on the knee stability - anterior-posterior translation, internal and external rotations after the double-bundle reconstruction of Anterior Cruciate Ligament and to compare the stability after single-bundle and double-bundle reconstruction using a computer navigation system.

DETAILED DESCRIPTION:
The purpose of this prospective study is to evaluate the influence of both bundles on the knee stability - anterior-posterior translation, internal and external rotations after the double-bundle reconstruction of Anterior Cruciate Ligament (ACL) and to compare the stability after single-bundle and double-bundle reconstruction using a computer navigation system.

Methods Anterior-posterior translation, internal rotation, and external rotation were recorded in the deficient condition (without ACL), in the anteromedial-reconstructed, posterolateral-reconstructed, and in the whole ACL-reconstructed condition for double-bundle reconstructions and before and after the ACL reconstruction in single-bundle group. KT-1000 was used to evaluate anterior-posterior translation.

ELIGIBILITY:
Inclusion Criteria:

* isolated ACL lesion and primary ACL replacement

Exclusion Criteria:

* replacement of ACL with navigation system

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
measurement of rotational and anterior-posterior movement tibia to femur before the replacement of ACL | one hour
  measurement of rotational and anterior-posterior movement tibia to femur before the replacement the ACL (single bundle)or after the tonisation of one portion of ACL in double bundle type of reconstruction of ACL in the operating sale

SECONDARY OUTCOMES:
measurement of rotational and anterior-posterior movement tibia to femur after the replacement of ACL | one hour
  measurement of rotational and anterior-posterior movement tibia to femur after the replacement the ACL (single bundle)or after the tonisation of second portion of ACL in double bundle type of reconstruction of ACL in the operating sale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Komzák, Principal Investigator — Hospital Znojmo
Locations (1):
- Hospital Znojmo, Znojmo, Czech Republic, Czechia

REFERENCES:
- See also: web page of investigator affiliation — http://nemzn.cz